CLINICAL TRIAL: NCT05414916
Title: Pain Relief Strategies for Dressing Change in Chronic Wounds: Qualitative Interview Stage
Brief Title: Pain Relief Strategies for Dressing Change in Chronic Wounds
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: 165104
Record Dates: First submitted 2022-05-25; First posted 2022-06-10 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-06

CONDITIONS: Pain; Chronic Wound
Keywords: Dressing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A small-scale study using interviews to explore patients', carers' and health care professionals' experience of pain relief strategies currently used in UK practice for dressing change in chronic wounds.

DETAILED DESCRIPTION:
In 2012/2013, the National Health Service (NHS) managed an estimated 2.2 million adults >18 years of age with a wound, of which 48% were estimated as being chronic. A chronic wound is an open sore in the skin that does not heal, or takes a long time to heal, and frequently comes back. Chronic wounds include pressure ulcers (bed sores), venous (vein-related) leg ulcers, and foot ulcers in people who have diabetes. Pain is a common experience for people living with chronic wounds and can result from the wound itself, treatments for chronic wounds, including dressing changes; or be anticipatory. Pain during dressing change has been reported as the worst part of living with chronic wounds, followed closely by wound cleansing. Furthermore, dried out dressings and adherent products are most likely to cause pain and trauma at dressing changes as is gauze, while products such as hydrogels and soft silicone dressings are least likely. Evidence suggests that supporting the surrounding skin during dressing removal is not considered a priority, despite evidence that many adhesive products may lead to skin stripping and potential skin trauma and pain.

There is at present little recent evidence of pain relief strategies that are currently being used in the UK for dressing change in chronic wounds that includes patients', carers' and healthcare professionals' (people who work in the NHS) use and experience of these. This qualitative research will explore providers' and recipients' self-reported experiences of chronic wound care, and explore strategies used to reduce pain at dressing change. It will ask about the perceived success of these strategies from different participant perspectives, along with how pain is assessed. Perceptions of what factors might contribute to pain at dressing change (e.g., dressing and wound type, skill levels) will be captured along with perceptions of what could improve the management of pain at dressing change.

ELIGIBILITY:
Inclusion Criteria:

* Living with a chronic wound, informally or privately caring for someone with a chronic wound or providing medical care (e.g. dressing change) for someone with a chronic wound
* Ability to give informed consent
* Aged aged 18 years or above

Exclusion Criteria:

* Vulnerable patients (e.g. severe mental illness, learning difficulties, dementia, care home residents)
* Inability to provide informed consent
* Inability to communicate in English
* Not living with a chronic wound, informally or privately caring for someone with a chronic wound or providing medical care (e.g. dressing change) for someone with a chronic wound
* Under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients registered with a GP practice in England who are living with a chronic wound, informal or private carers for people living with a chronic wound and health care professionals (staff nurses, tissue viability specialists) providing primary or secondary medical care for someone with a chronic wound.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To identify what strategies have been used by patients, carers and healthcare professionals to reduce or remove pain associated with dressing changes in chronic wounds. | 6 months
  experiences and strategies will be explored and captured from qualitative data collected from semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cooper, PhD, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Goole Health Centre, Goole, Yorkshire
  - Clifton Medical Centre, Rotherham, Yorkshire

IPD SHARING:
Plan to Share IPD: No